CLINICAL TRIAL: NCT06368466
Title: A Prospective Cross-Sectional Study to Evaluate Diagnostic Sensitivity and Specificity of iStatis HBsAg Test at the Point-Of-Care Sites
Brief Title: A Study to Evaluate Diagnostic Sensitivity and Specificity of iStatis HBsAg Test at the Point-Of-Care Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Collaborators: St Vincent's Hospital Melbourne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: CLS-016A
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis B; Hepatitis B Infection
Keywords: Hepatitis B rapid test; Hepatitis B infection; Hepatitis B iStatis test; Hepatitis B point of care test
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iStatis Performance (Experimental): capillary (fingerstick) blood, EDTA venous whole blood, serum and plasma samples will be tested on iStatis HBsAg Test
  Interventions: Device: iStatis HBsAg Test
- Reference Test to evaluate iStatis Performance (No Intervention): Either serum or plasma samples will undergo reference lab testing using DiaSorin Liaison XL Murex HBsAg Quant Assay and DiaSorin Murex HBsAg Confirmatory assay

INTERVENTIONS:
Device: iStatis HBsAg Test — capillary (fingerstick) blood, EDTA venous whole blood, serum and plasma samples are tested on the iStatis HBsAg Test
  Arms: iStatis Performance

SUMMARY:
A prospective cross-sectional study in which surgically non-invasive sample-taking is done only for the purpose of the study. Capillary (fingerstick) whole blood and EDTA venipuncture whole blood are collected by a healthcare professional. The collected samples of capillary and EDTA whole blood are tested on iStatis and EDTA whole blood sample will be processed to obtain serum and plasma samples to be tested on the iStatis. An aliquot of the collected serum sample will be shipped to the central laboratory for confirmatory testing. The results from iStatis HBsAg Test results will not be used for patient management decisions.

DETAILED DESCRIPTION:
From each enrolled patient, a total of 2 different blood samples (capillary and venous whole blood) will be collected, processed, and categorized under the following categories:

- Sample 1: 50μL of Capillary (fingerstick) (see section 8.6.2) Sample 2: 16ml of Venous whole blood (further extraction of serum, and plasma samples) (see section 8.6.2) Sample 1 consisting of capillary (fingerstick) and Sample 2 venous whole blood sample will be tested on iStatis HBsAg Test on site according to the 'Test Procedure' described in the Instructions for Use (IFU) supplied with the reagents. Sample 2 containing of 1 EDTA and SST venous whole blood samples will be separately processed to obtain plasma and serum samples, respectively, and will be tested onsite on the iStatis. An aliquot of the serum sample stored and frozen at -20ᵒC at the testing site will be transferred to the central laboratory to establish further reference testing. Upon arrival of the sample, it will undergo an initial test using DiaSorin Liaison XL Murex HBsAg Quant Assay, REF. [310250] following the IFU of this reference assay. If the first run of the assay yields a "non-reactive/Negative" result, it will be reported as such. However, if the sample is "Reactive/Positive" in the first run of the assay testing, it will be retested on the same assay in duplicate, following the manufacturer's instructions. A final "Reactive/Positive" result means that at least one of the duplicate repeat tests was reactive, if neither of the duplicate repeat tests yields a reactive results, the final report in the DiaSorin Liaison XL Murex HBsAg Quant Assay requires three tests to confirm. Samples with a reportable "Reactive/Positive" result in the DiaSorin Liaison XL Murex HBsAg Quant Assay will undergo further testing using DiaSorin Murex HBsAg Confirmatory assay, REF. [9F80-01]. A "Reactive/Positive" result in this test will confirm the presence of the relevant marker.

ELIGIBILITY:
Inclusion Criteria:

* Patients/subjects (males, females, and pregnant women) getting tested for HBV for one or more of the following reasons:

  * at risk for HBV
  * having signs and symptoms indicative of HBV
  * pregnant and have HBV.
  * Re-infected with HBV (previously positive)
* Patients/subjects of 18 years or older and, who are able to give/sign the informed consent.

Exclusion Criteria:

* Patient younger than 18 years old
* Patients unable to provide written informed consent.
* Patients currently undergoing treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Performance | 3 Months
  To evaluate the performance of the iStatis HBsAg POC test with the RT-PCR test at the point of care sites by a healthcare professional.
Sensitivity and Specificity | 3 Months
  To assess the sensitivity and specificity of the iStatis HBsAg POC test with four different sample types.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Melbourne, Melbourne, Fitzroy Victoria, Australia

IPD SHARING:
Plan to Share IPD: No